CLINICAL TRIAL: NCT03234023
Title: A Remote Nursing-Guided Secondary Prevention Programme in Acute Coronary Syndrome. The SPRING Randomized Controlled Trial
Brief Title: Secondary PRevention in Cardiovascular Disease by a Nursing Guided Program (SPRING)
Acronym: SPRING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital A Coruña (Other)
Responsible Party: Principal Investigator, CARMEN NERI FERNANDEZ POMBO, Research Nurse., University Hospital A Coruña
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017/101; SPRING (Other: University Hospital A Coruña)
Record Dates: First submitted 2017-07-25; First posted 2017-07-31 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Acute Coronary Syndrome; Nutrition; Physical Activity; Secondary Prevention
MeSH Terms: conditions — Acute Coronary Syndrome; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INTERVENTION GROUP (Active Comparator): The participants of this group will follow recommendations of food, physical exercise, control of consumption of drugs and consumption of alcohol and tobacco.
  Interventions: Behavioral: INTERVENTION GROUP
- CONTROL GROUP (No Intervention): The participants of this group are submitted to the standard intervention.

INTERVENTIONS:
Behavioral: INTERVENTION GROUP — Offer recommendations of healthy living habits and control of pharmacy administration
  Arms: INTERVENTION GROUP

SUMMARY:
DESIGN: Controlled clinical trial with single randomization, unmasked, open and multicentric.

CENTERS: University Hospital of A Coruña and University Hospital of Ferrol CONDITION TO STUDY: Acute Coronary Syndrome (ACS). INTERVENTION:monitored outhospital not inhospital supervised. MAIN OBJECTIVE: To determine the incidence of major adverse events (total mortality, new ACS, coronary revascularization, all-cause hospitalization) during the one-year period after hospitalization for ACS.

DETAILED DESCRIPTION:
The SPRING study aims to learn whether a remote, nurse-guided secondary prevention program reduces adverse events in patients who suffer an infarction during the subsequent one-year period. The SPRING study focuses not only on adverse events but also on the patients' state of life in terms of diet, physical exercise, emotional state, tobacco use, and adherence to medical treatment. Nursing is a profession in charge of preserving the health of patients, which is why the remote secondary cardiovascular prevention program of this study is coordinated by a nurse.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have suffered an ACS in the health area of A Coruña or Ferrol from the beginning of the study inclusion period until reaching the fixed sample size.
* Ages between 18 and 75 years.
* Patients with ability to read and understand the participation sheet in the study.
* Patients signing informed consent to participate in the study.
* Patients living in the health care area of HUAC or HUF.

Exclusion Criteria:

* Patients who are dependent for the Basic Activities of Daily Living (BADL) or who suffer from severe cognitive impairment (which makes reliable anamnesis impossible).
* Patients with a Left Ventricular Ejection Fraction (LVEF) less than or equal to 35%.
* Patients with a NYHA III / IV score and / or the Canadian Cardiovascular Association (CCS) scale of IV.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 484 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2023-02-05 (Actual); Study Completion 2023-02-05 (Actual)

PRIMARY OUTCOMES:
major adverse events | 1 year
  total mortality, new ACS, coronary revascularization, hospitalization for any cause

SECONDARY OUTCOMES:
cardiovascular mortality | 1 year
  cardiovascular mortality
cardiovascular hospitalization | one year
  cardiovascular hospitalization
stroke | 1 year
  stroke
tobacco | 1 year
  questionnaire
physical activity | 1 year
  mets
nutrition | 1 year
  mediterranean diet
emotion state | 1 year
  questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Neri Fernández Pombo, PhD, Principal Investigator — University Hospital A Coruña; Guillermo Aldama López, MD, Principal Investigator — University Hospital A Coruña; José Manuel Vázquez Rodríguez, MD, Principal Investigator — University Hospital A Coruña; Raquel Marzoa Rivas, MD, Principal Investigator — University Hospital Ferrol; Manuel López Pérez, MD, Principal Investigator — University Hospital Ferrol; Marta Lorenzo Carpente, Nurse, Principal Investigator — University Hospital Ferrol; Jose Angel Rodriguez Fernández, MD, Principal Investigator — University Hospital A Coruña
Locations (2):
- Spain (2):
  - University Hospital of Ferrol, Ferrol, A Coruña
  - University Hospital of A Coruña, A Coruña, Galicia

IPD SHARING:
Plan to Share IPD: No
The data of the participants can not be used by other researchers

REFERENCES:
- [Derived] Fernandez-Pombo CN, Aldama-Lopez G, Lorenzo-Carpente M, Lopez-Perez M, Marzoa-Rivas R, Rodriguez-Fernandez JA, Vazquez-Rodriguez JM. A Remote Nursing-Guided Secondary Prevention Programme in Acute Coronary Syndrome. The SPRING Randomised Controlled Trial. J Adv Nurs. 2026 Feb;82(2):1803-1818. doi: 10.1111/jan.17046. Epub 2025 May 15. PMID 40372009